CLINICAL TRIAL: NCT01087827
Title: Anatomical Determinants of Forearm and Upper Arm Oscillometric Blood Pressure Differences
Brief Title: Body Structures Determining Differences in Forearm and Upper Arm Blood Pressures
Status: Completed | Type: Observational
Sponsor: Christiana Care Health Services (Other)
Collaborators: University of Delaware (Other)
Responsible Party: Sponsor
Other Study IDs: CCC29150; NURS175154 (Other: University of Delaware IRB)
Record Dates: First submitted 2010-03-08; First posted 2010-03-16 (Estimated); Last update posted 2012-11-07 (Estimated); Status verified 2012-11

CONDITIONS: Blood Pressure
Keywords: oscillometric blood pressure; cuff site; forearm blood pressure; upper arm blood pressure; anthropometric measurements; tonometry; site of blood pressure measurement; measurement accuracy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The first purpose of this study is to see how blood pressures taken at different sites, specifically the forearm, upper arm and heart vessels, are different. The second purpose is to see if body structures such as vessel size and depth, size of the arm, and amount of tissue in the arm influence differences in blood pressures taken at these sites. The third purpose is to develop a mathematical model of the waves generated by the arm arteries (brachial and radial) to predict differences in forearm and upper arm blood pressures. The results of the study may be used to design more accurate non-invasive blood pressure monitors for the forearm site.

DETAILED DESCRIPTION:
Accurate blood pressure (BP) measurement is required to provide appropriate healthcare. Inaccurate BPs may lead to under and/or over-treatment of health conditions and medical diseases such as hypertension. Blood pressure (BP) measurement using automatic, non-invasive oscillometric monitors is common in clinics, physicians'offices and hospital settings. The brachial (upper arm) site is the gold standard for non-invasive BPs. However, in some situations, this site is inaccessible due to injury, surgery, dialysis shunts, intravenous devices, and lymphedema. When the upper arm is difficult to access or the available BP cuffs do not fit an individual's arm, the forearm site is often the preferable alternative. The increased incidence of obesity nationally also contributes to the heightened use of forearm BPs. Questions remain concerning the accuracy of forearm non-invasive BP measurements. Although most researchers report that upper arm and forearm readings are not interchangeable, size of differences vary for individuals and factors influencing differences in readings have not been thoroughly investigated.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age
* able to speak and write in English

Exclusion Criteria:

* Individuals with non-intact skin where the BP cuffs would be placed
* Individuals with injury or surgery to the arm within the last month
* Individuals with lymphedema in the limb selected for measurements
* Individuals with arteriovenous fistulas
* Individuals with differences > 5 mm Hg between right and left arm oscillometric systolic BP measurements
* Individuals with documented valvular disease
* Individuals with atrial fibrillation or atrial flutter (as recommended by BP device manufacturers due to device inaccuracy)
* Individuals with an International Normalized Ratio (INR) > 1.7
* Individuals with intravenous catheters in both arms
* Individuals who require immediate cardiac surgery or unanticipated emergency treatment or who are unstable during the procedure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients undergoing non-emergent cardiac catheterization
Sampling Method: Non-Probability Sample
Enrollment: 51 (Actual)
Dates: Start 2010-03; Primary Completion 2012-03 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
anatomical determinants of forearm and upper arm blood pressure differences | 6 months
  body mass index, upper arm circumference, biceps skin-fold measurement, forearm and upper arm vessel diameter, forearm and upper arm vessel depth

SECONDARY OUTCOMES:
blood pressure differences; quantitative model of waveform propagation and reflection able to predict differences between upper arm and forearm blood pressures | 6 months
  blood pressure at forearm, upper arm, aortic root
  radial artery tonometry to determine radial artery waveform and pressure measurements non-invasively

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen A Schell, PhD, Principal Investigator — University of Delaware
Locations (1):
- Christiana Hospital, Newark, Delaware, United States

REFERENCES:
- [Background] Schell K, Lyons D, Bradley E, Bucher L, Seckel M, Wakai S, Carson E, Waterhouse J, Chichester M, Bartell D, Foraker T, Simpson EK. Clinical comparison of automatic, noninvasive measurements of blood pressure in the forearm and upper arm with the patient supine or with the head of the bed raised 45 degrees: a follow-up study. Am J Crit Care. 2006 Mar;15(2):196-205. PMID 16501139
- [Background] Schell K, Bradley E, Bucher L, Seckel M, Lyons D, Wakai S, Bartell D, Carson E, Chichester M, Foraker T, Simpson K. Clinical comparison of automatic, noninvasive measurements of blood pressure in the forearm and upper arm. Am J Crit Care. 2005 May;14(3):232-41. PMID 15840897
- [Background] Schell K, Morse K, Waterhouse JK. Forearm and upper-arm oscillometric blood pressure comparison in acutely ill adults. West J Nurs Res. 2010 Apr;32(3):322-40. doi: 10.1177/0193945909351887. PMID 20581399
- [Background] Schell K, Waterhouse,JK. Comparison of forearm and upper arm automatic noninvasive blood pressures in college students. Internet Journal of Advanced Nursing Practice 2007, 9 (1): 10 pages
- [Background] Schell KA, Richards JG, Farquhar WB. The effects of anatomical structures on adult forearm and upper arm noninvasive blood pressures. Blood Press Monit. 2007 Feb;12(1):17-22. doi: 10.1097/MBP.0b013e3280858cd0. PMID 17303983
- [Background] Rose WC, Johnson DA, Spaeth JR, Edwards J, Beris, AN. Computational and experimental investigation of arterial hemodynamics. Proc. 2008 Int. Mech. Eng. Conf. Exp. Boston: ASME, 2008; 1-8.